CLINICAL TRIAL: NCT06051487
Title: Evaluation of the Effect of Titanium Dioxide Nanoparticles Addition to Acrylic Baseplates of Orthodontic Functional Appliances
Brief Title: Evaluation of Anti Bacterial Effect of Titanium Dioxide Nanoparticles on Baseplates of Twin Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dentist
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Gingival Inflammation
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium dioxide nanoparticles containing group (Other): participants using twin block appliance in which titanium dioxide nanoparticles added to acrylic baseplates to evaluate its antibacterial effect
  Interventions: Other: titanium dioxide nanoparticles in test group
- control (Other): participants use twin block appliance without any addition to acrylic base plates
  Interventions: Other: titanium dioxide nanoparticles in test group

INTERVENTIONS:
Other: titanium dioxide nanoparticles in test group — Titanium dioxide nanoparticles added to acrylic baseplate in test group

SUMMARY:
Background The objective of this study was to evaluate the antibacterial effect of Titanium dioxide nanoparticles incorporated into the acrylic baseplates of maxillary part of twin block appliances in orthodontic patients during the treatment period.

Material and methods Twenty-six patients were selected randomly and divided into two groups(n=13). Test group patients were used orthodontic functional appliances containing Titanium dioxide nanoparticles in acrylic baseplates. Control group patients were used orthodontic functional appliances without Titanium dioxide nanoparticles in acrylic baseplates. Swap samples were taken from palatal gingiva facing fitting surface of acrylic component of maxillary part of twin block appliance for each patient at five times intervals (base line sample, after one, two, four, and six months) then cultured in blood agar plates to calculate bacterial colony count.

DETAILED DESCRIPTION:
Design of the appliance

For all of the chosen patients, the Twin Block, which consists of upper and lower bite blocks, was constructed. In this study the upper bite block was used. The upper part incorporates labial bow with U loop around canines and Adam clasps on the upper first molars for retention. Midline screw may be added to the upper part of the appliance to aid in the correction of the posterior cross bite if occurred during treatment.

Appliance construction (dental laboratory step) Based on cast models of each patient, acrylic baseplates for orthodontic appliances were manufactured using auto-polymerizing PMMA resin, the monomer-to-polymer ratio recommended by the manufacturer, and standard acrylization, trimming, and finishing-polishing processes The acrylic material used for fabrication of the appliance was (Acrostone acrylic material, under exclusive liscence, England). The manufacturer's suggested powder-liquid volume ratio is 3:1 representing 22 g of the polymer and 10 mL of the liquid monomer. Powder-liquid volume ratio for construction of appliance was calculated . This created samples were the control group.

Intervention Titanium dioxide nano powder was prepared at City of Scientific Research and Technological Applications (SRTA-City) in Egypt.

During the appliance containing TiO2 nanoparticles construction, first of all, the calculated quantity of titanium dioxide nano powder was mixed manually with acrylic resin polymer for 60 s by shaking the powders inside a small container and subsequently, the calculated quantity of the monomer was added to obtain a PMMA containing TiO2 NPs .This created samples were the test group. the powder was mixed with the liquid as recommended by the manufacturer, applied to a mold and ﬂasked. Then the acrylic baseplate was finished and polished.

Clinical step:

The patients were instructed to use the device (twin block) full-time, including while they slept. The patients were instructed not to use mouthwashes, antibiotics, or xylitol products during this time but to continue brushing their teeth as usual and eating a normal diet instead. Prior to sample collection, the patients were told not to brush their teeth or practise other oral hygiene routines for 24 hours, and they were also told not to eat or drink for an hour.

Sample:

Swap Samples were taken just before wearing the appliance (base line sample) then at the following time intervals of wearing appliance for each group (after one month, after two-months, after four-months, and after six months).

Swap was taken from palatal gingiva facing fitting surface of acrylic baseplate of maxillary part of twin block appliance for each patient using sterilized cotton swap then placed in 1ml of broth solution in sterilized tube.

Broth solution (thioglycolate broth) which act as transport media used to refresh bacteria if it present and preserve it until send to lab.

Sample examination (laboratory step) Sample examination was done in Microbiology Diagnostics and Infection Control unit (MDICU), Medical Microbiology and Immunology Department, Faculty of Medicine, Mansoura University.

After sample had been send to the lab, vortex was done for it using Vortex Mixer VM-300 Gemmy for one or two minute to release all sample from the swap in the solution(1ml). Then swap was discarded and broth solution was used. We used 10 microns of the solution. it was cultured in blood agar plate. Solution was placed on the top of the plate using swap, descended on vertical line in the middle part of the plate then horizontal lines passing through this vertical line then the plate was placed in the incubator for 24 hours to calculate the colony forming unit / ml for streptococcus mutans.

ELIGIBILITY:
Inclusion Criteria:

* early permanent dentition (ages 9 to 14)
* mandibular retrusion-related class II skeletal deformity
* overjet more than 4mm

Exclusion Criteria:

* systemic diseases
* congenital craniofacial deformity
* inflammatory or infectious diseases within the previous month
* taking medication in the last month, such as fluoride or antibiotics
* frequent consumers of sorbitol- and xylitol-containing products
* mouth rinses
* unusual or specific dietary habits
* cleft lip or palate
* unusual habits or previous orthodontic treatment.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Bacterial colony count | samples was taken within five time intervals (base line samples, at one month, at two months, at four months, at six months)
  Changes in bacterial colony count under acrylic base plate in Participants using twin block appliance containing titanium dioxide nanoparticles in comparison to participant using appliance not containing titanium dioxide nanoparticles

CONTACTS AND LOCATIONS:
Overall Officials: Ghada M Elabd, Principal Investigator — Master degree student
Locations (1):
- Mansoura university, Al Mansurah, Egypt